CLINICAL TRIAL: NCT04666974
Title: Delivering Online Cognitive Behavioural Therapy (iCBT) to Address Mental Health Challenges in Correctional Officers and Other Public Safety Personnel
Brief Title: Delivering ICBT to Address Mental Health Challenges in Correctional Officers and Other Public Safety Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Nazanin Alavi (Other)
Collaborators: Online PsychoTherapy Clinic (Other)
Responsible Party: Sponsor-Investigator, Dr. Nazanin Alavi, Assistant Professor, Principle Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSIY-684-20
Record Dates: First submitted 2020-12-05; First posted 2020-12-14 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Mental Health Issue; Anxiety Disorders; Depressive Disorder; Post-Traumatic Stress Disorder
Keywords: Clinical; Population Health; Correctional Workers; Online Psychotherapy; Mental Health Issues; Online Cognitive Behavioural Therapy
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants in Phase 3 will be randomly assigned to either iCBT + Treatment as Usual or just Treatment as Usual. In phase 4, participants will be randomly assigned to either iCBT + Treatment as Usual or in-person CBT + Treatment as Usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase 3: iCBT + Treatment As Usual (Experimental): CWs in the iCBT group, will be assigned to one the six therapy modules, based on their gender and diagnosis (i.e. Female/Male * GAD, MDD or PTSD). Each CW will be assigned a specific clinician (a trained psychiatrist/psychologist/ social worker) who would be their care liaison through the study. Each week, the clinician would send one session of the 12-session curriculum to the CW on a pre-determined day of the week. Each weekly session consists of 20-30 slides followed by a homework assignment. It usually takes 40-60 minutes for a participant to complete one weekly session which they have to complete by a specific day of the week. The clinician will review the CW's assignments and provide feedback on their performance. The clinician feedback is structured and takes approximately 15 minutes to complete. The clinician will then send the content for the next session along with the feedback.
  Interventions: Behavioral: iCBT
- Phase 3: Treatment as Usual (No Intervention): Participants will complete clincally validated questionnaires to measure symptoms while continuing with their regular daily activities and treatments (if any) (i.e., exercise, diet, medications, etc.)
- Phase 4: iCBT + Treatment as Usual (Experimental): Participants will be randomly assigned to this group and take part in the iCBT module program from phase 3.
  Interventions: Behavioral: iCBT
- Phase 4: In-Person CBT + Treatment as Usual (Active Comparator): Participants will be randomly assigned to this group and complete in-person CBT with similar content, homework, and feedback as in the iCBT + TAU group. All in-person CBT will be delivered by a trained professional and each session will take approximately 60-75 minutes.
  Interventions: Behavioral: In-Person CBT

INTERVENTIONS:
Behavioral: iCBT — Online CBT modules will be completed weekly with content mirroring in-person CBT for their diagnosis. Homework will be submitted weekly through the OPTT platform which will be reviewed by a trained professional who will provide personalized feedback.
  Arms: Phase 3: iCBT + Treatment As Usual; Phase 4: iCBT + Treatment as Usual
Behavioral: In-Person CBT — Participants will be assigned to in-person CBT that will mirror the content and homework covered in the iCBT group. It will be delivered by professionals and attended weekly.
  Arms: Phase 4: In-Person CBT + Treatment as Usual

SUMMARY:
Public safety personnel (PSP) have regular and often intense exposure to potentially traumatic events at work and are at higher risk for developing mental health problems such as posttraumatic stress disorder (PTSD). Studies have shown up to 4 times higher suicidal ideation, attempt and death among this population compared to the general population. Despite the high rate of mental health problems among PSPs, their willingness to receive mental healthcare support is fairly low, mainly due to the stigma attached to these disorders. Those who are willing to seek help face unique barriers including their irregular shift hours, limiting their access to resources otherwise available to the public. Given these challenges and the critical contribution of PSPs to public safety, developing innovative solutions to address their mental health must be a healthcare priority.

This proposal aims to study the efficacy of using an innovative approach in delivering mental health online, to address mental health problems among correctional workers (CW), who are especially prone to mental health problems given the high rate of workplace violence. It is hypothesized that using an online platform to deliver cognitive behavioural therapy (CBT), would lower the stigma of receiving care in a secure and confidential environment, easing CW's concerns about stigma from co-workers. The content is delivered through interactive and engaging therapy modules, designed for specific groups of CWs and customized by situational examples to make therapy more relatable. These online modules would provide CWs with 24/7 access to therapy content, solving the irregular work hour problem. The online CBT modules developed in this study would provide high quality and clinically validated resources to address mental health problems of CWs all across Canada. Knowledge acquired through this project could also be beneficial to using iCBT in general for addressing mental health challenges among other PSPs.

DETAILED DESCRIPTION:
Phase 1 An expert end-user group of correctional workers (n = 5) will help the research team across all phases of this project. These experts will have in-depth knowledge of CW problems and will be chosen in consultation with CW union members. Provincial correctional workers (n = 40) (20 male & 20 female) will be recruited to participate in individual interviews and then in virtual focus groups through Microsoft Teams. These interviews will be used to identify the main mental health challenges and the best methods to address them in the context of different groups of CWs (administrative, operational workers, direct vs indirect contact with prisoners, working in a prison vs working in probation offices, etc.) and investigate the barriers specific to each group. Interview/focus group members will be recruited through flyers (distributed in place of work), advertisements in specialized journals, through union representatives and through word of mouth. Each individual will be independently interviewed by a trained research assistant (RA) hired for the project (60-90-minute interviews). Interviews will occur remotely via a secure video conference with Microsoft Teams. Questions will include topics of the level of interaction with prisoners, types and frequency of violence at work, sexual assault, work condition (staffing, shift length, relationship with superiors and co-workers, work-load, over-crowdedness), socio-economic factors (racial, gender, language, sexuality, religious discrimination), mental challenges (anxiety, depression, PTSD, suicidal ideation), resources (training, peer-support and professional help) and frequency they use them, reasons for refraining to use resources, the preferred method of support (onsite vs offsite, individual vs. group), and attitude towards online care (willing to do so and what content they want to be covered). Information gathered through individual interviews will form the basis for further virtual focus group discussions with Microsoft Teams. The final format of the questionnaire will be decided in consultation between the PI and all co-applicants including experts of the field (Drs. Simpson, Gerritsen and Martin) and the expert end-user group to ensure the validity of each question from psychiatric, epidemiologic, psychologic, forensic and professional aspects.

Following individual interviews, 5 half-day focus groups (8 participants per group, 2 exclusively female, 2 exclusively male, 1 evenly mixed) will be conducted to gather more information regarding issues uncovered in individual interviews. These focus groups will occur remotely via a virtual video conference with Microsoft Teams. A list of challenges to be addressed in phases 2-4 will be formed from these interviews. The PI, one psychiatrist, one psychologist, one RA and at least 2 members of the end-user expert group will attend each group meeting to form a better understanding of the problems faced by each group. All interviews and focus group discussions will be recorded and transcribed verbatim for further discussion at the investigative team meetings.

Phase 2 Following the first round of content development, each CBT module will be presented to the end-user expert group and a smaller number of interview/focus group participants (10 males & 10 females) for feedback. Each participant will be asked to provide feedback on one of the six therapeutic modules regarding content, form, presentation, examples and helpfulness, based on the challenges it tries to address. All feedback will be summarized and compiled by project RAs and discussed in 6 separate focus group discussions attended by the PI, one psychiatrist, one psychologist, one RA and at least 2 members of the end-user expert group. Each participant is requested to attend two virtual focus group discussions on the module they have not seen yet or commented on. This step is done to ensure each participant can provide feedback on all gender-specific therapy contents A list of recommended changes to each module is developed through these group discussions. Recommendations will be reviewed by the PI, co-applicants and the knowledge users for clinical validation. The final changes, compiled by clinicians, will be applied to each module and proper graphical changes will be made.

Phase 3 CW participants will be recruited for this phase of the study through flyers (distributed in place of work), advertisements in specialized journals, through union representatives and through word of mouth. Also, in this phase, the investigators will accept participants based on referrals from family physicians or psychiatrists in small cities with correctional facilities who could be easily informed of the study through academic recourses. All CWs will go through a comprehensive initial mental health assessment by a psychiatrist either in person or through video, using Ontario Telemedicine Network (OTN). All diagnoses are validated by a structured Mini-International Neuropsychiatric Interview (MINI) performed by a trained RA. To be included for the study, the CW should be between 18-55 years of age at the start of the study, diagnosed with either major depressive disorder (MDD), generalized anxiety disorder (GAD), or post-traumatic stress disorder (PTSD) according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) by a psychiatrist on the team, competence to provide informed consent and participate, able to speak and read English, and consistent and reliable access to the internet. The CWs are excluded from the study if they are diagnosed with hypomanic/manic episodes, psychosis, severe alcohol or substance use disorder, and active suicidal or homicidal ideation.

The 100 CWs (50 males, 50 females) meeting the inclusion/exclusion criteria will complete a set of socioeconomic and demographic questionnaires and baseline quantitative clinical questionnaires delivered online through the Online Psychotherapy Tool (OPTT) (DASS42, Q-LES-Q, QIDS-SR16, PHQ-9, GAD7, PCL-5). OPTT is a secure, cloud-based, online platform. After the initial assessment, the CWs will be randomly assigned to one of two study arms; 50 CWs receiving iCBT + TAU (treatment) vs 50 CWs receiving TAU (control).

CWs in the iCBT group will be assigned to one of the six therapy modules, based on their gender and diagnosis (i.e. Female/Male * GAD, MDD or PTSD). Each CW will be assigned a specific clinician (a trained psychiatrist/psychologist/ social worker) who would be their care liaison through the study. Each week, the clinician would send one session of the 12-session curriculum to the CW on a pre-determined day of the week. Each weekly session consists of 20-30 slides followed by a homework assignment. It usually takes 40-60 minutes for a participant to complete one weekly session which they have to complete by a specific day of the week. The clinician will review the CW's assignments and provide feedback on their performance. The clinician feedback is structured and takes approximately 15 minutes to complete. The clinician will then send the content for the next session along with the feedback.

CWs in both study arms will be asked to complete biweekly questionnaires depending on diagnosis to evaluate any change in diagnostic symptoms. At the end of week 12, the CWs will be asked to complete a final set of questionnaires (same as baseline) and another MINI. In order to evaluate long-term effects, follow up evaluations of both study arms will be done at 6 and 12 months following initial enrolment using the same quantitative questionnaires. In addition to clinical evaluations, CWs receiving iCBT will fill a qualitative questionnaire regarding their experience using OPTT. These questions will include -whether OPTT was aesthetically appealing, whether OPTT was intuitive, if they needed technical support, whether the navigation was simple enough, devices they used to access their therapy. The results of this feasibility survey will be discussed with the end-user expert group and system changes will be made for a better experience for the next phase. As data is collected through the experiment, anonymized data (diagnosis, initial and week 12 assessments, bi-weekly progress and 6- and 12-month follow-up assessments) will be shared with the other co-investigators to use in publications or presentations.

Phase 4 CWs will be recruited for the study using the same methods as in phase 3, going through a comprehensive interview by a psychiatrist, and validated by a MINI performed by trained RAs. Similar inclusion/exclusion criteria as in phase 3 are used for this phase as well. 100 CWs (gender-balanced) meeting inclusion/exclusion criteria will complete a set of socio-economic and demographic questionnaires and baseline quantitative clinical questionnaires delivered online through OPTT. Following the initial assessment, the CWs will then be randomly assigned to either iCBT + TAU (n=50) or in-person CBT + TAU (n=50).

CWs in either study arm will be will then be assigned to one of the therapy modules, based on primary diagnosis and gender (Female/Male * GAD, MDD or PTSD). Each CW will be assigned a specific clinician (trained psychiatrist/psychologist/social worker) who will be their care liaison through the study. The in-person CBT group will receive similar content, homework, and feedback as in the iCBT group. All in-person CBT will be delivered by a trained professional (psychiatrist/psychologist/SW). Each appointment is expected to take 60-75 minutes per week.

CWs in both study arms will complete biweekly tests depending on diagnosis to evaluate progress. At the end of the 12 weeks, the CWs will be asked to complete a final set of quantitative questionnaires and to complete another MINI. Feasibility questionnaires will be sent to CWs in the iCBT group and the responses will be discussed with the end-user expert group to form recommendations for improving OPTT. As data is collected through the study, anonymized data (diagnosis, initial, bi-weekly and 12-week assessments) will be openly shared for other researchers to use as well.

ELIGIBILITY:
Inclusion Criteria:

* Correctional worker or public safety personnel
* Diagnosis of either Major Depressive Disorder, Generalized Anxiety Disorder, or Post-Traumatic Stress Disorder
* Competence to provide informed consent and participate
* Speak and read English
* Consistent and reliable access to the internet

Exclusion Criteria:

* Diagnosis of hypomanic/manic episodes
* Psychosis
* Severe alcohol or substance abuse disorder
* Active suicidal or homicidal ideation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Symptoms (Depression and Anxiety Scale - DASS 42 Item) | Baseline, week 2, 4, 6, 8, 10, 12, 6-month follow-up, 12-month follow-up
  Questionnaire for symptomlogy changes. Scale of 0-3, 3 is worse.
Change in Symptoms (Quality of Life Enjoyment and Satisfaction - Q-LES-Q) | Baseline, week 2, 4, 6, 8, 10, 12, 6-month follow-up, 12-month follow-up
  Questionnaire for symptomlogy changes. Scale of 0-5, 5 is best
Change in Symptoms (Quick Inventory of Depressive Symptoms Self Report - QIDS-SR 16 Item) | Baseline, week 2, 4, 6, 8, 10, 12, 6-month follow-up, 12-month follow-up
  Questionnaire for symptomlogy changes. Scale of 0-3, 3 is worse.
Change in Symptoms (Patient Health Questionnaire - PHQ 9 Item) | Baseline, week 2, 4, 6, 8, 10, 12, 6-month follow-up, 12-month follow-up
  Questionnaire for symptomlogy changes. Scale of 0-3. 3 is worse.
Change in Symptoms (Generalized Anxiety Disorder - GAD 7) | Baseline, week 2, 4, 6, 8, 10, 12, 6-month follow-up, 12-month follow-up
  Questionnaire for symptomlogy changes. Scale of 0-3, 3 is worse.
Change in Symptoms (PTSD Checklist - PCL-5) | Baseline, week 2, 4, 6, 8, 10, 12, 6-month follow-up, 12-month follow-up
  Questionnaire for symptomlogy changes. Scale of 0-4, 4 is worse.

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin Alavi, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Alavi N, Stephenson C, Omrani M, Gerritsen C, Martin MS, Knyahnytskyi A, Zhu Y, Kumar A, Jagayat J, Shirazi A, Moghimi E, Patel C, Knyahnytska Y, Simpson AIF, Zaheer J, Andersen J, Munshi A, Groll D. Delivering an Online Cognitive Behavioral Therapy Program to Address Mental Health Challenges Faced by Correctional Workers and Other Public Safety Personnel: Protocol for a Mixed Methods Study. JMIR Res Protoc. 2021 Jul 22;10(7):e30845. doi: 10.2196/30845. PMID 34088656